CLINICAL TRIAL: NCT01362608
Title: A Randomized, Double-blind, Double-dummy, Active Controlled Study of Canakinumab (ACZ885) on the Treatment and Prevention of Gout Flares in Patients With Frequent Flares for Whom NSAIDs and/ or Colchicine Are Contraindicated, Not Tolerated or Ineffective
Brief Title: Safety & Efficacy of Canakinumab (ACZ885) in Patients With Frequent Flares for Whom Nonsterodial Anti-Inflammatory Drug (NSAIDs) and/ or Colchicine Are Contraindicated, Not Tolerated or Ineffective
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CACZ885H2358; 2010-024172-26
Record Dates: First submitted 2011-05-24; First posted 2011-05-30 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Gouty Arthritis
Keywords: Gout; Inflammatory gout; acute gout
MeSH Terms: conditions — Arthritis, Gouty; Gout | interventions — canakinumab; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Canakinumab and placebo matching to triamcinolone acetonide (Experimental): ACZ885H
  Interventions: Drug: Canakinumab, ACZ885
- Triamcinolone acetonide 40 mg (Active Comparator): ACZ885H
  Interventions: Drug: Triamcinolone acetonide

INTERVENTIONS:
Drug: Canakinumab, ACZ885 — Canakinumab and placebo matching to triamcinolone acetonide
  Arms: Canakinumab and placebo matching to triamcinolone acetonide
Drug: Triamcinolone acetonide — Triamcinolone acetonide 40 mg and placebo matching to canakinumab
  Arms: Triamcinolone acetonide 40 mg

SUMMARY:
The purpose of this pivotal Phase III study is to support the registration of canakinumab for the indication of gout in China, a replicate of global studies CACZ885H2356 & CACZ885H2357 by demonstrating in patients with frequent flares of gout for whom NSAIDs and/or colchicine are contraindicated, not tolerated or ineffective, canakinumab 150 mg s.c. given upon acute gout flares relieves the signs and symptoms and prevents recurrence of gout flares compared to triamcinolone acetonide 40 mg i.m.

ELIGIBILITY:
Inclusion criteria:

* Meeting diagnosis criteria for acute arthritis of primary gout.
* Start of acute gout flare within 5 days prior to study visit 1
* History of ≥ 3 gout flares within the 12 months prior to study start
* Evidence of contraindication (absolute or relative), or intolerance, or lack of efficacy for either NSAIDs and/or colchicines

Exclusion criteria:

* Requirement for administration of antibiotics against latent tuberculosis (TB), e.g., isoniazide
* Refractory heart failure (Stage D).
* Unstable cardiac arrhythmias or unstable symptomatic coronary ischemia
* Secondary gout, chemotherapy induced gout, lead induced gout and transplant gout
* Rheumatoid arthritis, evidence/suspicion of infectious/septic arthritis, or other acute inflammatory arthritis

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2011-06-20 (Actual); Primary Completion 2015-05-19 (Actual); Study Completion 2015-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- Novartis Investigative Site, Ciudad Autonoma de Bs As, Argentina
- China (10):
  - Novartis Investigative Site, Hefei, Anhui
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Wuhan
- Poland (3):
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Wroclaw
- Novartis Investigative Site, Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Groups:
- ACZ885 150 mg: Patients were treated with canakinumab 150 mg s.c and matching placebo for triamcinolone acetonide i.m.
- Triamcinolone Acetonide 40 mg: triamcinolone acetonide 40 mg i.m. and matching placebo for canakinumab s.c.
Period: Overall Study
Arm/Group | ACZ885 150 mg | Triamcinolone Acetonide 40 mg
Started | 67 | 69
Completed | 63 | 61
Not Completed | 4 | 8
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACZ885 150 mg | Triamcinolone Acetonide 40 mg | Total
Number analyzed (Participants) | 67 | 69 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 66 | 124
  >=65 years | 9 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (11.98) | 49.2 (11.37) | 49.7 (11.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 66 | 67 | 133

OUTCOME MEASURES:

1. Primary Outcome: The Change in the Gout Pain Intensity in the Target Joint Following ACZ885 Administration Measured by Visual Analog Scale (VAS)
Description: A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in postsurgical patients (knee replacement, hysterectomy, or laparoscopic myomectomy) who described their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0 - 4 mm), mild pain (5- 44 mm), moderate pain (45-74 mm), and severe pain (75- 100 mm)
Time Frame: at 72 hours post-dose
Population: Full Analysis set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACZ885 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 67 | 69
units on a scale | 18.2 (3.03) | 37.9 (3.03)
Statistical Analysis 1: Comparison: ACZ885 150 mg vs Triamcinolone Acetonide 40 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -19.69, 95% CI 2-sided [-28.2 to -11.2]

2. Primary Outcome: Time to First New Flare: Survival Analysis by Treatment: Kaplan Meier Analysis
Description: Measure canakinumab 150 mg s.c. is superior to triamcinolone acetonide 40 mg i.m. with respect to the time to the first new gout flare in observation period of 12 weeks
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | ACZ885 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 67 | 69
Participants | 5 (3.03) [1.19 to 13.93] | 17 (3.03) [15.29 to 36.71]
Statistical Analysis 1: Comparison: ACZ885 150 mg vs Triamcinolone Acetonide 40 mg; Test type: Superiority or Other; p = 0.0043, Regression, Cox; Hazard Ratio (HR) = 0.26, 95% CI 2-sided [0.10 to 0.71]

3. Secondary Outcome: The Number of Patients With at Least 1 New Gout Flare
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | ACZ885 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 67 | 69
participants
  1 new flare | 3 | 15
  2 new flares | 0 | 1
  3 new flares | 0 | 0
  > 3 new flares | 2 | 1

4. Secondary Outcome: Patients Assessment of Gout Pain Intensity in the Most Effected Joint (0-100mm VAS): Summary Statistics by Timepoint and Treatment
Description: as for outcome 1
Time Frame: baseline through 12 weeks
Population: Full Analysis set
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | ACZ885 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 67 | 69
unit on a scale
  baseline | 72.3 (13.18) | 74.5 (12.88)
  6 hours post-dose | 53.0 (22.06) | 58.8 (23.83)
  12 hours post-dose | 41.7 (19.56) | 51.8 (27.07)
  24 hours post-dose | 30.9 (18.23) | 48.6 (29.13)
  48 hours post-dose | 22.0 (18.64) | 43.9 (30.69)
  72 hours post-dose | 17.4 (17.02) | 36.6 (30.62)
  7 days post-dose | 10.1 (15.61) | 24.0 (27.31)
  4 weeks post-dose | 9.5 (17.25) | 17.9 (25.31)
  8 weeks post-dose | 6.8 (13.64) | 16.0 (24.24)
  12 weeks post-dose | 6.8 (12.92) | 13.0 (19.77)

5. Secondary Outcome: Patient's Assessment of Gout Pain Intensity in the Most Affected Joint (Likert Scale): Frequency Table by Timepoint and Treatment
Description: Patients will score their current pain intensity in the most affected joint of the gout flare on a 5-point Likert scale (none, mild, moderate, severe, extreme).
Time Frame: baseline through week 12
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | ACZ885 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 67 | 69
participants
  baseline none | 0 | 0
  baseline mild | 2 | 3
  baseline moderate | 25 | 18
  baseline severe | 37 | 44
  baseline extreme | 3 | 4
  6 hours post-dose none | 0 | 0
  6 hours post-dose mild | 18 | 14
  6 hours post-dose moderate | 28 | 26
  6 hours post-dose severe | 17 | 29
  6 hours post-dose extreme | 2 | 0
  12 hours post-dose none | 1 | 2
  12 hours post-dose mild | 28 | 19
  12 hours post-dose moderate | 28 | 26
  12 hours post-dose severe | 7 | 21
  12 hours post-dose extreme | 1 | 1
  24 hours post-dose none | 3 | 4
  24 hours post-dose mild | 40 | 20
  24 hours post-dose moderate | 19 | 25
  24 hours post-dose severe | 2 | 20
  24 hours post-dose extreme | 1 | 0
  48 hours post-dose none | 10 | 10
  48 hours post-dose mild | 48 | 21
  48 hours post-dose moderate | 7 | 20
  48 hours post-dose severe | 2 | 14
  48 hours post-dose extreme | 0 | 2
  72 hours post-dose none | 14 | 12
  72 hours post-dose mild | 45 | 26
  72 hours post-dose moderate | 8 | 16
  72 hours post-dose severe | 0 | 9
  72 hours post-dose extreme | 0 | 4
  4 days post-dose none | 21 | 14
  4 days post-dose mild | 39 | 29
  4 days post-dose moderate | 7 | 13
  4 days post-dose severe | 0 | 10
  4 days post-dose extreme | 0 | 0
  7 days post-dose none | 32 | 23
  7 days post-dose mild | 29 | 25
  7 days post-dose moderate | 5 | 10
  7 days post-dose severe | 1 | 8
  7 days post-dose extreme | 0 | 0
  4 weeks post-dose none | 43 | 24
  4 weeks post-dose mild | 17 | 25
  4 weeks post-dose moderate | 4 | 6
  4 weeks post-dose severe | 1 | 0
  4 weeks post-dose extreme | 0 | 0
  8 weeks post-dose none | 39 | 30
  8 weeks post-dose mild | 22 | 21
  8 weeks post-dose moderate | 2 | 6
  8 weeks post-dose severe | 2 | 2
  8 weeks post-dose extreme | 0 | 0
  12 weeks post-dose none | 41 | 25
  12 weeks post-dose mild | 18 | 28
  12 weeks post-dose moderate | 3 | 8
  12 weeks post-dose severe | 2 | 1
  12 weeks post-dose extreme | 0 | 1

6. Secondary Outcome: Patient's Global Assessment of Response to Treatment: Frequency Table by Timepoint and Treatment Using a Likert Scale.
Description: Patients will score their response to pain on a 7-point Likert scale (excellent, good ,acceptable, slight,poor,very poor,not done).
Time Frame: 72 hours through week 12
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | ACZ885 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 67 | 69
participants
  72 hours post-dose excellent | 7 | 3
  72 hours post-dose good | 40 | 17
  72 hours post-dose acceptable | 14 | 18
  72 hours post-dose slight | 4 | 11
  72 hours post-dose poor | 1 | 10
  72 hours post-dose very poor | 0 | 0
  72 hours post-dose not done | 0 | 1
  7 days post-dose excellent | 16 | 4
  7 days post-dose good | 38 | 20
  7 days post-dose acceptable | 9 | 18
  7 days post-dose slight | 1 | 7
  7 days post-dose poor | 1 | 16
  7 days post-dose very poor | 0 | 0
  7 days post-dose not done | 0 | 1
  4 weeks post-dose excellent | 15 | 6
  4 weeks post-dose good | 33 | 19
  4 weeks post-dose acceptable | 13 | 14
  4 weeks post-dose slight | 4 | 7
  4 weeks post-dose poor | 0 | 9
  4 weeks post-dose very poor | 0 | 0
  4 weeks post-dose not done | 0 | 2
  8 weeks post-dose excellent | 18 | 8
  8 weeks post-dose good | 35 | 16
  8 weeks post-dose acceptable | 10 | 18
  8 weeks post-dose slight | 2 | 9
  8 weeks post-dose poor | 0 | 8
  8 weeks post-dose very poor | 0 | 0
  8 weeks post-dose not done | 0 | 1
  12 weeks post-dose excellent | 16 | 4
  12 weeks post-dose good | 37 | 21
  12 weeks post-dose acceptable | 10 | 21
  12 weeks post-dose slight | 0 | 7
  12 weeks post-dose poor | 1 | 9
  12 weeks post-dose very poor | 0 | 0
  12 weeks post-dose not done | 3 | 3

7. Secondary Outcome: Physician's Assessment of Tenderness: Frequency Table by Timepoint and Treatment
Description: Physicians will score their response to pain on a 5-point Likert scale (no pain, pain,pain and winces,pain winces and withdraws and not assessed).
Time Frame: baseline 72 hours,7 days 4 weeks, 8 weeks and 12 weeks post dose
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | ACZ885 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 67 | 69
participants
  Baseline no pain | 0 | 0
  Baseline pain | 15 | 16
  Baseline pain and winces | 31 | 29
  Baseline pain, winces and withdraws | 21 | 24
  Baseline not assessed | 0 | 0
  72 hours post-dose no pain | 23 | 16
  72 hours post-dose pain | 37 | 26
  72 hours post-dose pain and winces | 5 | 11
  72 hours post-dose pain, winces and withdraws | 1 | 3
  72 hours post-dose not assessed | 0 | 0
  7 days post-dose no pain | 41 | 26
  7 days post-dose pain | 23 | 27
  7 days post-dose pain and winces | 2 | 10
  7 days post-dose pain , winces and withdraws | 0 | 2
  7 days post-dose not assessed | 0 | 0
  4 weeks post-dose no pain | 54 | 30
  4 weeks post-dose pain | 10 | 19
  4 weeks post-dose pain and winces | 1 | 3
  4 weeks post-dose pain, winces and withdraws | 0 | 3
  4 weeks post-dose not assessed | 0 | 0
  8 weeks post-dose no pain | 54 | 38
  8 weeks post-dose pain | 11 | 19
  8 weeks post-dose pain and winces | 0 | 1
  8 weeks post-dose pain winces and withdraws | 0 | 1
  8 weeks post-dose not assessed | 0 | 0
  12 weeks post-dose no pain | 53 | 39
  12 weeks post-dose pain | 7 | 22
  12 weeks post-dose pain and winces | 2 | 1
  12 weeks post-dose pain, winces and withdraws | 2 | 0
  12 weeks post-dose not assessed | 0 | 0

8. Secondary Outcome: Physician's Assessment of Swelling: Frequency Table by Timepoint and Treatment
Description: as for outcome 7
Time Frame: baseline 72 hours,7 days 4 weeks, 8 weeks and 12 weeks post dose
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | ACZ885 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 67 | 69
participants
  Baseline No swelling | 1 | 3
  Baseline Palpable | 13 | 12
  Baseline Visible | 29 | 39
  Baseline Bulging beyond the joint margins | 24 | 15
  Baseline not assessed | 0 | 0
  72 hours post-dose No swelling | 38 | 22
  72 hours post-dose Palpable | 15 | 15
  72 hours post-dose Visible | 12 | 18
  72 hrs post-dose Bulging beyond the joint margins | 1 | 1
  72 hours post-dose not assessed | 0 | 0
  7 days post-dose No swelling | 53 | 35
  7 days post-dose Palpable | 9 | 18
  7 days post-dose Visible | 3 | 9
  7 days post-dose Bulging beyond the joint margins | 1 | 3
  7 days post-dose not assessed0 | 0 | 0
  4 weeks post-dose No swelling | 60 | 40
  4 weeks post-dose Palpable | 2 | 9
  4 weeks post-dose Visible | 3 | 4
  4 weeks post-dose Bulging beyond the joint margins | 0 | 2
  4 weeks post-dose not assessed | 0 | 0
  8 weeks post-dose No swelling | 63 | 49
  8 weeks post-dose Palpable | 0 | 6
  8 weeks post-dose Visible | 2 | 4
  8 weeks post-dose Bulging beyond the joint margins | 0 | 0
  8 weeks post-dose not assessed | 0 | 0
  12 weeks post-dose No swelling | 61 | 52
  12 weeks post-dose Palpable | 1 | 6
  12 weeks post-dose Visible | 2 | 2
  12 wks post-dose Bulging beyond the joint margins | 0 | 2
  12 weeks post-dose not assessed | 0 | 0

9. Secondary Outcome: Physician's Assessment of Erythema: Frequency Table by Timepoint and Treatment
Description: Physicians will score their response of erythema on a 4-point Likert scale (absent, present not assessed and not assessable).
Time Frame: baseline 72 hours,7 days 4 weeks, 8 weeks and 12 weeks post dose
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | ACZ885 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 67 | 69
participants
  Baseline Absent | 19 | 19
  Baseline present | 48 | 50
  Baseline not assessed | 0 | 0
  Baseline not assessable | 0 | 0
  72 hours post-dose absent | 54 | 41
  72 hours post-dose present | 11 | 15
  72 hours post-dose not assessed | 0 | 0
  72 hrs post-dose not assessable | 1 | 0
  7 days post-dose absent | 62 | 57
  7 days post-dose present | 3 | 8
  7 days post-dose not assessed | 0 | 0
  7 days post-dose not assessable | 1 | 0
  4 weeks post-dose absent | 63 | 49
  4 weeks post-dose present | 1 | 6
  4 weeks post-dose not assessed | 0 | 0
  4 weeks post-dose not assessable | 1 | 0
  8 weeks post-dose absent | 65 | 56
  8 weeks post-dose present | 0 | 3
  8 weeks post-dose not assessed | 0 | 0
  8 weeks post-dose not assessable | 0 | 0
  12 weeks post-dose absent | 62 | 61
  12 weeks post-dose present | 1 | 1
  12 weeks post-dose not assessed | 0 | 0
  12 wks post-dose not assessable | 1 | 0

10. Secondary Outcome: Physician's Assessment of Range of Motion: Frequency Table by Timepoint and Treatment
Description: Physicians will score their response ofrange of motion on a 5-point Likert scale (normal,mildly restricted, moderately restricted, severely restricted and immolbilized).
Time Frame: baseline through week 12
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | ACZ885 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 67 | 69
participants
  baseline normal | 0 | 0
  baseline mildly restricted | 3 | 6
  baseline moderately restricted | 32 | 24
  baseline severely restricted | 27 | 39
  baseline immobilzed | 5 | 0
  72 hours post-dose normal | 20 | 15
  72 hours post-dose mildly restricted | 33 | 19
  72 hours post-dose moderately restricted | 11 | 14
  72 hours post-dose severely restricted | 2 | 7
  72 hours post-dose immobilized | 0 | 1
  7 days post-dose normal | 35 | 26
  7 days post-dose mildly restricted | 25 | 20
  7 days post-dose moderately restricted | 4 | 15
  7 days post-dose severely restricted | 1 | 3
  7 days post-dose immobilized | 0 | 1
  4 weeks post-dose normal | 49 | 25
  4 weeks post-dose mildly restricted | 12 | 22
  4 weeks post-dose moderately restricted | 3 | 7
  4 weeks post-dose severely restricted | 1 | 1
  4 weeks post-dose immobilized | 0 | 0
  8 weeks post-dose normal | 51 | 32
  8 weeks post-dose mildly restricted | 12 | 18
  8 weeks post-dose moderately restricted | 1 | 6
  8 weeks post-dose severely restricted | 1 | 3
  8 weeks post-dose immobilized | 0 | 0
  12 weeks post-dose normal | 50 | 30
  12 weeks post-dose mildly restrcted | 1 | 23
  12 weeks post-dose moderately restricted | 2 | 6
  12 weeks post-dose severely restricted | 1 | 3
  12 weeks post-dose immobilized | 0 | 0

11. Secondary Outcome: Time to at Least a 50% Reduction in Baseline Pain Intensity: Survival Analysis by Treatment
Description: Kaplan Meier estimate
Time Frame: 12 weeks
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | ACZ885 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 67 | 69
hours | 24.0 [24.0 to 48.0] | 48.0 [24.0 to 72.0]

12. Secondary Outcome: Time to Complete Resolution of Pain: Survival Analysis by Treatment
Description: Kaplan Meier estimate
Time Frame: 12 weeks
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | ACZ885 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 67 | 69
hours | 168.0 [120.0 to 168.0] | 168.0 [NA to NA] — CI cannot calculated for this parameter as it is "too narrow to exist". The CI limits are time points where events happened or censored. When we decrease the confidence level from 99% to 95%, no observed time point meets the criterion.

13. Secondary Outcome: Time to First Rescue Medication Intake
Time Frame: 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ACZ885 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 67 | 69
hours | 31.8 (30.45) | 41.5 (38.8)

14. Secondary Outcome: Percent Patients Who Took Rescue Medication
Time Frame: 12 weeks
Population: FAS
Measure: Number; unit: percentage
Arm/Group | ACZ885 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 67 | 69
percentage
  Baseline flare (n= 29,42) | 43.3 | 60.9
  Last post-baseline flare (n=3,4) | 75.0 | 44.4

15. Secondary Outcome: Amount of Rescue Medication Taken at Baseline Flare and Post Baseline Flare.
Description: Paracetamol / acetaminophen, Prednisolone and Prednisone taken at baseline flare and post baseline flare.
Time Frame: 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | ACZ885 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 67 | 69
mg
  Baseline flare Paracetamol / acetaminophen | 342.5 (680.53) | 451.4 (744.19)
  Baseline flare Prednisolol | 1.1 (4.25) | 5.0 (15.29)
  Baseline Flare Prednisone | 0.7 (5.52) | 5.2 (30.42)
  Baseline flare Codeine | 0.0 (0.00) | 0.4 (3.61)
  Last post-baseline flare Paraceta/acetamin n=4,9 | 287.5 (337.58) | 222.2 (666.67)
  Last post-baseline flare Prednisolone n=4,9 | 5.0 (10.00) | 4.4 (8.82)
  Last post-baseline flare Prednisone n=4,9 | 0.0 (0.00) | 0.6 (1.67)

16. Secondary Outcome: High Sensitivity C-reactive Protein [hsCRP] Measured in the Serum at 72 Hours Post Dose
Time Frame: 72 hours post dose
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | ACZ885 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 67 | 69
mg/L | 5.5 [4.4 to 6.9] | 7.2 [5.7 to 9.2]

ADVERSE EVENTS:
Groups:
- ACZ885 150mg sc: ACZ885 150mg sc
- Triam 40mg im: Triam 40mg im
Arm/Group | ACZ885 150mg sc | Triam 40mg im
Serious Adverse Events (participants affected / at risk) | 0/67 | 1/69
Other Adverse Events (participants affected / at risk) | 0/67 | 4/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACZ885 150mg sc (N=67) | Triam 40mg im (N=69)
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACZ885 150mg sc (N=67) | Triam 40mg im (N=69)
Hypertension (Vascular disorders) | 0 | 4

LIMITATIONS AND CAVEATS:
This study was terminated early. The decision to terminate study was not out of concerns for efficacy or safety of canakinumab

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.